CLINICAL TRIAL: NCT03369704
Title: A 12 Week, Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Omalizumab in Adult and Adolescent Patients With Inadequately Controlled Severe Japanese Cedar Pollinosis Despite the Current Recommended Therapies
Brief Title: Study of Efficacy and Safety of Omalizumab in Severe Japanese Cedar Pollinosis Adult and Adolescent Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIGE025F1301
Record Dates: First submitted 2017-11-14; First posted 2017-12-12 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: cryptomeria, omalizumab, seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omalizumab (Experimental): Eligible patients randomized to this arm received omalizumab subcutaneously for 12 weeks
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): Eligible patients randomized to this arm received placebo subcutaneously for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab were administered by subcutaneous injection. Dose (75 to 600 mg) and dosing frequency (every 2 or 4 weeks) were determined by serum total IgE level (IU/mL) and body weight (kg) measured at the screening epoch according the dosing table.
  Arms: Omalizumab
Drug: Placebo — Placebo were administered by subcutaneous injection. Dose (75 to 600 mg) and dosing frequency (every 2 or 4 weeks) were determined by serum total IgE level (IU/mL) and body weight (kg) measured at the screening epoch according the dosing table.
  Arms: Placebo

SUMMARY:
The purpose of this study was to demonstrate the efficacy and safety of omalizumab compared with placebo, on top of SoC (anti-histamine and nasal corticosteroid) in adult and adolescent patients with severe Japanese cedar pollinosis, whose symptoms were inadequately controlled despite the current recommended therapies (nasal corticosteroids plus one or more medications out of anti-histamine, leukotriene receptor antagonist, or prostaglandin D2/thromboxane A2 receptor antagonist) in the previous 2 Japanese cedar pollen seasons.

ELIGIBILITY:
Inclusion criteria:

* A clinical history of Japanese cedar pollinosis defined by the following

  * Took nasal corticosteroid plus one or more medications out of antihistamine (second generation), leukotriene receptor antagonist, or prostaglandin D2 thromboxane A2 receptor antagonist in Japanese cedar pollen seasons in 2016 and 2017.
  * Had inadequately controlled symptoms of Japanese cedar pollinosis lasting at least one week in the Japanese cedar pollen season in 2017 despite the nasal corticosteroid plus one or more medications out of anti-histamine (second generation), leukotriene receptor antagonist, or prostaglandin D2/thromboxane A2 receptor antagonist (regardless of having perennial allergic rhinitis or not)
* Serum cedar pollen-specific Immunoglobulin E (IgE) levels of ≥ score of 3 by CAP/RAST-FEIA, ImmunoCAP or MAST at the screening epoch.
* Developing a symptom of Japanese cedar pollinosis during the period from first observational day in cedar pollen in Kanto area to initial drug administration (Visit 101), as defined by the following

  * Having any nasal or ocular symptom (≥ score of 1 in sneezing, rhinorrhea, nasal congestion, itchy eye or watery eye) in at least 2 days or
  * Having both any nasal symptom (≥ score of 1 in sneezing, rhinorrhea, nasal congestion) and any eye symptom (≥ score of 1 in itchy eye or watery eye) in at least one day, which is confirmed by patient e-diary (unless a symptom is clearly consider to take place due to other than Japanese cedar pollinosis/allergic rhinitis (e.g., upper respiratory tract infection, or common cold)).
* Body weight and serum total IgE level at screen epoch within the dosing table range; body weight of ≥ 20 to ≤ 150 kg and serum total IgE levels of ≥ 30 to ≤ 1500 IU/mL at a maximum.

Exclusion Criteria:

* With an active rhinitis other than allergic rhinitis (e.g acute or chronic rhinitis, idiopathic rhinitis).
* With an active nose disease other than allergic rhinitis (e.g., acute or chronic rhinosinusitis or deflected septum) which is expected to affect the evaluation of efficacy of the study drug judged by the investigator.
* With elevated serum IgE levels for reasons other than allergy (e.g., parasite infections, hyperimmunoglobulin E syndrome, Wiskott-Aldrich Syndrome or clinical allergic bronchopulmonary aspergillosis).
* With a severe asthma treated with high dose inhaled corticosteroid (≥ 800 μg/day fluticasone propionate or an equivalent for aged ≥ 16 to <75 years, > 200 μg/day for aged ≥ 12 to <16 years).
* Who are receiving operative treatment for allergic rhinitis (e.g., electrocoagulation, laser surgery, 80% trichloroacetic acid chemo-surgery, inferior turbinectomy or posterior nasal neurectomy) within 1 years prior to the screening epoch.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Japan (18):
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Urayasu, Chiba
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Arakawa-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Nakano-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Toshima-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=429
- See also: A Pediatric Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 22 centers in Kanto-area of Japan.
Pre-assignment Details: 337 patients were randomized
Groups:
- Omalizumab: Omalizumab administered subcutaneously for 12 weeks
- Placebo: Placebo administered subcutaneously for 12 weeks
Period: Treatment Epoch
Arm/Group | Omalizumab | Placebo
Started | 162 | 175
Completed | 158 | 172
Not Completed | 4 | 3
Not completed — technical problems | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Adverse Event | 2 | 0
Period: Follow-up Epoch
Arm/Group | Omalizumab | Placebo
Started | 161 | 174
Completed | 160 | 174
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set (RAN): The RAN included all randomized patients, regardless of whether they received any study drug. Patients in the RAN was analyzed according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 162 | 175 | 337
Age, Customized [Number; unit: Participants]
  < 15 years | 4 | 6 | 10
  15 <=, < 65 years | 149 | 158 | 307
  >= 65 years | 9 | 11 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 97 | 196
  Male | 63 | 78 | 141
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 162 | 175 | 337

OUTCOME MEASURES:

1. Primary Outcome: Mean Nasal Symptom Score
Description: Nasal symptoms (sneezing, rhinorrhea and nasal congestion) were recorded by the patient everyday in their e-Diary, on a scale of 0 (none) to 4 (intense/severe). Nasal symptom score (0-12 point) consisted of score for severity of sneezing (0-4 point), rhinorrhea (0-4 point) and nasal congestion (0-4 point).
  Severe symptom period: The three weeks where the cumulative value of the mean daily nasal symptom score is the maximum. The three weeks must also meet one of the following criteria: 2) ≥ 70% of the period with concomitant use of fluticasone propionate is included in this three weeks. 2) ≥ 70% of this three weeks includes the period with concomitant use of fluticasone propionate. If not, severe symptom period was extended at a minimum to meet one of the criteria above. The severe symptom period will be defined as: the three weeks where the cumulative value of the mean daily nasal symptom score will be the maximum.
Time Frame: Severe symptom period (from 23Feb2018 to 24March2018)
Population: Full analysis set (FAS): The FAS consisted of all patients in the RAN who received at least 1 dose of study drug. Among patients in the FAS, those who had nasal symptom scores for at least 50% of days during the severe symptom period were included.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
score | 3.66 (0.151) | 4.69 (0.144)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; p < 0.001, ANCOVA — H0: Omalizumab is not different to placebo with respect to mean nasal symptom score over the severe symptom period. H1: Omalizumab is different to placebo with respect to mean nasal symptom score over the severe symptom period; Least Square Mean = -1.03, 95% CI 2-sided [-1.44 to -0.62], Standard Error of Mean 0.209 — nasal symptom score

2. Secondary Outcome: Mean Ocular Symptom Score and Mean Nasal Ocular Symptom Score
Description: Ocular symptoms (itchy and watery eye) were recorded by the patient everyday in their e-Diary, on a scale of 0 (none) to 4 (intense/severe). Ocular symptom score (0-8 point) consisted of score for severity of itchy eye (0-4 point) and watery eye (0-4 point).
  Nasal ocular symptom score consisted of nasal symptom score and ocular symptom score.
  Nasal ocular symptom score is the sum of nasal symptom score (0-12) and ocular symptom score (0-8) 0 presents no nasal ocular symptom and 20 presents worse outcome.
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
Score
  Mean ocular symptom score | 2.45 (0.115) | 3.32 (0.110)
  Mean nasal ocular symptom score | 6.11 (0.240) | 8.01 (0.228)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -1.89, 95% CI 2-sided [-2.55 to -1.24], Standard Error of Mean 0.331 — Nasal Ocular Symptom
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.87, 95% CI 2-sided [-1.18 to -0.55], Standard Error of Mean 0.159 — Ocular symptom

3. Secondary Outcome: Mean Nasal Symptom Medication Score, Mean Ocular Symptom Medication Score, and Mean Nasal Ocular Symptom Medication Score
Description: Medication scores were given for fluticasone propionate (nasal, 2 point), fexofenadine hydrochloride (oral, 1 point), tramazoline hydrochloride (nasal, 1 point), and levocabastine hydrochloride (ocular, 1 point). Symptom medication score consisted of severe symptom period.
  Nasal symptom medication score is the sum of nasal symptom score and medication score (fexofenadine hydrochloride, fluticasone propionate, tramazoline hydrochloride) Ocular symptom medication score is the sum of ocular symptom score and medication score (fexofenadine hydrochloride, levocabastine hydrochloride) Nasal ocular symptom medication score is the sum of nasal symptom score, ocular symptom score and medication score (fexofenadine hydrochloride, fluticasone propionate, tramazoline hydrochloride, levocabastine hydrochloride).
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
score
  Mean nasal symptom medication score | 6.19 (0.166) | 7.29 (0.158)
  Mean ocular symptom medication score | 3.91 (0.137) | 4.86 (0.130)
  Mean nasal ocular symptom medication score | 9.10 (0.271) | 11.15 (0.259)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -1.10, 95% CI 2-sided [-1.55 to -0.64], Standard Error of Mean 0.229 — nasal symptom medication score
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.95, 95% CI 2-sided [-1.32 to -0.58], Standard Error of Mean 0.189 — ocular symptom medication score
Statistical Analysis 3: Comparison: Omalizumab; Test type: Other; ANCOVA = -2.05, 95% CI 2-sided [-2.78 to -1.31], Standard Error of Mean 0.375 — nasal ocular symptom medication score

4. Secondary Outcome: Mean Score for Severity of Sneezing, Rhinorrhea and Nasal Congestion
Description: Symptoms of sneezing, rhinorrhea and nasal congestion were evaluated on a scale of 0 (none) to 4 (intense/severe).
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
score
  Mean sneezing score | 1.15 (0.053) | 1.56 (0.050)
  Mean rhinorrhea score | 1.46 (0.063) | 1.79 (0.060)
  Mean nasal congestion score | 1.05 (0.058) | 1.34 (0.056)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.40, 95% CI 2-sided [-0.54 to -0.26], Standard Error of Mean 0.073 — sneezing score
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.34, 95% CI 2-sided [-0.51 to -0.16], Standard Error of Mean 0.088 — rhinorrhea score
Statistical Analysis 3: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.29, 95% CI 2-sided [-0.45 to -0.13], Standard Error of Mean 0.081 — nasal congestion score

5. Secondary Outcome: Mean Score for Severity of Itchy and Watery Eye
Description: Symptoms of itchy and watery eye were evaluated on a scale of 0 (none) to 4 (intense/severe).
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
score
  Mean itchy eye score | 1.47 (0.061) | 1.94 (0.058)
  Mean watery eye score | 0.98 (0.063) | 1.38 (0.060)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.47, 95% CI 2-sided [-0.63 to -0.30], Standard Error of Mean 0.084 — itchy eye score
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.40, 95% CI 2-sided [-0.57 to -0.23], Standard Error of Mean 0.087 — watery eye score

6. Secondary Outcome: Mean Score for Impairment of Daily Activities
Description: Impairment of daily activities were evaluated on a scale of 0 (none) to 4 (intense/severe).
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
score | 1.09 (0.052) | 1.43 (0.050)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.34, 95% CI 2-sided [-0.48 to -0.20], Standard Error of Mean 0.072 — score for impairment of daily activities

7. Secondary Outcome: Number of Symptom Free Days
Description: Nasal symptom free days (days with all nasal symptoms are not more than mild in severity) during the severe symptom period. Ocular symptom free days (days with all ocular symptoms are not more than mild in severity) during the severe symptom period.
Time Frame: Severe symptom period (from 23Feb2018 to 24March2018)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
days
  Nasal symptom free days | 15 [0 to 30] | 10 [0 to 30]
  Ocular symptom free days | 12 [0 to 30] | 6 [0 to 30]
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; p = 0.005, van Elteren test; Hodges-Lehmann Estimate = 3.0, 95% CI 2-sided [1.0 to 5.0], Standard Error of Mean 1.02 — Nasal symptom free days
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; p < 0.001, van Elteren test; Hodges-Lehmann Estimate = 4.0, 95% CI 2-sided [2.0 to 6.5], Standard Error of Mean 1.15 — Ocular symptom free days

8. Secondary Outcome: Completely Nasal Symptom Free Patients
Description: Completely nasal symptom free patients is the number of patients who were nasal symptom free (all nasal symptoms were not more than mild in severity) on all non-missing days and had nasal symptom scores for at least 26 days during the 30 days of severe symptom period.
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
Participants | 13 | 4
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; p = 0.005, logistic regression; Odds Ratio (OR) = 3.43, 95% CI 2-sided [1.21 to 9.75] — Completely nasal symptom free patients

9. Secondary Outcome: Rescue Medication Score
Description: Rescue medication scores were given for tramazoline hydrochloride (nasal, 1 point) and levocabastine hydrochloride (ocular, 1 point).
  Rescue medication score for nasal is medication score for Tramazoline hydrochloride, Rescue medication score for ocular is medication score for Levocabastine hydrochloride and Rescue medication score for nasal and ocular is the sum of medication score for Tramazoline hydrochloride and Levocabastine hydrochlorid
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
score
  Nasal rescue medication score | 0.20 (0.024) | 0.28 (0.023)
  Ocular rescue medication score | 0.46 (0.029) | 0.54 (0.027)
  Nasal ocular rescue medication score | 0.66 (0.045) | 0.82 (0.043)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.08, 95% CI 2-sided [-0.14 to -0.01], Standard Error of Mean 0.033 — Nasal rescue mediation score
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.08, 95% CI 2-sided [-0.16 to 0.00], Standard Error of Mean 0.040 — Ocular rescue medication score
Statistical Analysis 3: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.16, 95% CI 2-sided [-0.28 to -0.04], Standard Error of Mean 0.063 — Nasal ocular rescue medication score

10. Secondary Outcome: Rescue Medication Free Days
Description: Number of days with no rescue medication (tramazoline hydrochloride, levocabastine hydrochloride).
  Nasal ocular rescue medication free days were defined as the days with no use of tramazoline hydrochloride (nasal rescue medication) and levocabastine hydrochloride (ocular rescue medication).
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
days
  Nasal rescue medication free days | 27.0 [0 to 30] | 23.5 [0 to 30]
  Ocular rescue medication free days | 16.0 [0 to 30] | 11.0 [0 to 30]
  Nasal ocular rescue medication free days | 12.5 [0 to 30] | 9.0 [0 to 30]
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; p = 0.011, van Elteren test; Hodges-Lehmann Estimate = 1.5, 95% CI 2-sided [0.0 to 3.5], Standard Error of Mean 0.89 — Nasal rescue mediation free days
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; p = 0.074, van Elteren test; Hodges-Lehmann Estimate = 2.0, 95% CI 2-sided [0.0 to 4.8], Standard Error of Mean 1.21 — Ocular rescue medication free days
Statistical Analysis 3: Comparison: Omalizumab vs Placebo; Test type: Other; p = 0.098, van Elteren test; Hodges-Lehmann Estimate = 1.8, 95% CI 2-sided [0.0 to 4.0], Standard Error of Mean 1.02 — Nasal ocular rescue medication free days

11. Secondary Outcome: Number of Rescue Medication Used
Description: Amount number of rescue medication used (a total number of times used).
Time Frame: Severe symptom period (from 23Feb2018 to 24Mar2018)
Population: as for outcome 1
Measure: Median (Full Range); unit: Number of times used
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 158 | 174
Number of times used
  Number of rescue nasal medication used | 1.0 [0 to 120] | 6.0 [0 to 109]
  Number of ocular rescue medication used | 18.5 [0 to 109] | 28.5 [0 to 113]
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; p = 0.006, van Elteren test; Hodges-Lehmann Estimate = -2.0, 95% CI 2-sided [-4.5 to 0.0], Standard Error of Mean 1.15 — Nasal rescue mediation used
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; p = 0.012, van Elteren test; Hodges-Lehmann Estimate = -7.0, 95% CI 2-sided [-12.0 to -1.0], Standard Error of Mean 2.81 — Ocular rescue medication used

12. Secondary Outcome: Japanese Rhinoconjunctivitis Quality of Life Questionnaire (JRQLQ, No1) Score
Description: Nasal and eye symptoms (JRQLQ I) included 6 categories: Runny nose, Sneezing, Nasal congestion, Itchy nose, itchy eyes and watery eyes, on a 5-point scale of 0 to 4 (no symptoms to very severe symptoms). JRQLQ I score was a mean of these 6 categories. JRQLQ II included 17 items on a 5-point scale, 0 to 4 (no significant problem to very greatly). JRQLQ II scores was a mean of these 17 items. Overall face scale (JRQLQ III) evaluated overall symptoms, condition and feelings on a 5-point scale from 0 to 4 (fine to crying). Evaluation visit was defined as follows independently for each evaluation item and for each patient: 1) If there was a single visit during the severe symptom period, the visit was the evaluation visit. 2) If there were ≥ 2 visits during the severe symptom period and a) if Visit 105 was one of them, Visit 105 was the evaluation visit; b) if Visit 105 was outside the period, the closest visit to Visit 105 during the period was the evaluation visit.
Time Frame: Evaluation Visit, one visit during severe symptom period (23-Feb-2018 to 24-Mar-2018) for each patient
Population: Full analysis set (FAS): The FAS consisted of all patients in the RAN who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 160 | 175
Score
  Nasal and eye symptoms (JRQLQ I) | 1.27 (0.062) | 1.76 (0.059)
  Mean score of QoL-related questionnaire (JRQLQ II) | 0.70 (0.067) | 1.20 (0.064)
  Overall face scale (JRQLQ III) | 1.6 (0.08) | 2.2 (0.07)
Statistical Analysis 1: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.50, 95% CI 2-sided [-0.66 to -0.33], Standard Error of Mean 0.086 — JRQLQ I
Statistical Analysis 2: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.51, 95% CI 2-sided [-0.69 to -0.33], Standard Error of Mean 0.093 — JRQLQ II
Statistical Analysis 3: Comparison: Omalizumab vs Placebo; Test type: Other; ANCOVA = -0.6, 95% CI 2-sided [-0.8 to -0.4], Standard Error of Mean 0.10 — JRQLQ III

13. Secondary Outcome: Number of Participants With Anti-omalizumab Antibodes
Description: Number of participants with antibodies against the Fab and Fc region of omalizumab in serum.
Time Frame: Prior to first dosing (Day 1), At follow-up investigation which were conducted 20/22 weeks after 12 week-treatment epoch
Population: Safety set (SAF): The SAF consisted of all patients who received at least 1 dose of study drug. Patients in the SAF were analyzed according to treatment actually received.
Measure: Number; unit: participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 161 | 175
participants
  Anti-Fab-(pre-dose) | 0 | 0
  Anti-Fab (post dose): number analyzed (Participants) | 160 | 173
  Anti-Fab (post dose) | 0 | 0
  Anti-Fc-(pre-dose) | 1 | 2
  Anti-Fc-(post-dose): number analyzed (Participants) | 160 | 173
  Anti-Fc-(post-dose) | 0 | 2

14. Secondary Outcome: Serum Trough Omalizumab Concentration
Description: Blood samples were collected Prior to first dosing (Day 1), at Day 29, Day 57, Day 85 and follow-up investigation which were conducted 20/22 weeks after 12 week-treatment epoch
Time Frame: Prior to first dosing (Day 1), at Day 29, Day 57, Day 85 and 24 weeks after last dose
Population: Pharmacokinetic set (PK set): The PK set consisted of all randomized patients who received at least 1 dose of study drug and had at least 1 evaluable PK measurement. Patients in the PK set were analyzed according to the treatment they actually received.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Omalizumab
Number analyzed (Participants) | 161
μg/mL
  Day 1 (pre-dose) | 0 (0)
  Day 29: number analyzed (Participants) | 159
  Day 29 | 42.6 (34.8)
  Day 57: number analyzed (Participants) | 158
  Day 57 | 54.1 (42.3)
  Day 85 | 66.3 (49.0)
  Day 225/239: number analyzed (Participants) | 160
  Day 225/239 | 0.928 (1.11)

15. Secondary Outcome: Free IgE and Total IgE
Description: Blood samples were collected Prior to first dosing (Day 1), at Day 29, Day 57, Day 85 and follow-up investigation were conducted 20/22 weeks after 12 week-treatment epoch
Time Frame: Day 1, at Day 29, Day 57, Day 85 and 24 weeks after last dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 161 | 175
ng/mL
  Free IgE (Day 1 predose): number analyzed (Participants) | 52 | 54
  Free IgE (Day 1 predose) | NA (NA) — NA= Not Available. A result is NA when > 1/3 of the values were above ULOQ (upper limit of quantification). ULOQ defined as 150 ng/mL for free IgE | NA (NA) — NA= Not Available. A result is NA when > 1/3 of the values were above ULOQ (upper limit of quantification). ULOQ defined as 150 ng/mL for free IgE
  Free IgE (Day 29): number analyzed (Participants) | 159 | 62
  Free IgE (Day 29) | 21.3 (9.8) | NA (NA) — NA= Not Available. A result is NA when > 1/3 of the values were above ULOQ (upper limit of quantification). ULOQ defined as 150 ng/mL for free IgE
  Free IgE (Day 57): number analyzed (Participants) | 157 | 41
  Free IgE (Day 57) | 20.8 (10.1) | NA (NA) — NA= Not Available. A result is NA when > 1/3 of the values were above ULOQ (upper limit of quantification). ULOQ defined as 150 ng/mL for free IgE
  Free IgE (Day 85): number analyzed (Participants) | 161 | 39
  Free IgE (Day 85) | 18.6 (11.9) | NA (NA) — NA= Not Available. A result is NA when > 1/3 of the values were above ULOQ (upper limit of quantification). ULOQ defined as 150 ng/mL for free IgE
  Free IgE (Day 225/239): number analyzed (Participants) | 55 | 54
  Free IgE (Day 225/239) | NA (NA) — NA= Not Available. A result is NA when > 1/3 of the values were above ULOQ (upper limit of quantification). ULOQ defined as 150 ng/mL for free IgE | NA (NA) — NA= Not Available. A result is NA when > 1/3 of the values were above ULOQ (upper limit of quantification). ULOQ defined as 150 ng/mL for free IgE
  Total IgE (Day 1 pre-dose) | 524 (531) | 570 (641)
  Total IgE (Day 29): number analyzed (Participants) | 159 | 175
  Total IgE (Day 29) | 2040 (1620) | 558 (608)
  Total IgE (Day 57): number analyzed (Participants) | 158 | 173
  Total IgE (Day 57) | 2160 (1660) | 640 (721)
  Total IgE (Day 85) | 1960 (1480) | 673 (775)
  Total IgE (Day 225/239): number analyzed (Participants) | 160 | 173
  Total IgE (Day 225/239) | 702 (639) | 669 (783)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 85 days(end of the treatment epoch). Serious adverse events (SAE) were collected until 30 days after the end of the treatment epoch, up to approximately 4 months.
Description: Analysis was done in the safety set. n total 162 were randomized to IGE025 arm. 1 patient in IGE025 arm was randomized but received no study drug, so this patient was excluded from Safety set.
Groups:
- IGE025: Eligible patients randomized to this arm received omalizumab subcutaneously for 12 weeks
Arm/Group | IGE025 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/175
Serious Adverse Events (participants affected / at risk) | 1/161 | 0/175
Other Adverse Events (participants affected / at risk) | 26/161 | 21/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGE025 (N=161) | Placebo (N=175)
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGE025 (N=161) | Placebo (N=175)
Influenza (Infections and infestations) | 4 | 8
Nasopharyngitis (Infections and infestations) | 15 | 8
Pharyngitis (Infections and infestations) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT03369704/Prot_001.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT03369704/SAP_000.pdf